CLINICAL TRIAL: NCT02574273
Title: Pilot Trial of a Social Skills Group Treatment (Secret Agent Society Program) for Youth With Anxiety, ADHD, or Autistic Disorder
Brief Title: Pilot Trial of a Social Skills Group Treatment (Secret Agent Society Program)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1503015990
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Attention Deficit Hyperactivity Disorder (ADHD); Autistic Spectrum Disorder (ASD)
MeSH Terms: conditions — Anxiety Disorders; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secret Agent Society (SAS) Program (Active Comparator): The Secret Agent Society (SAS) Program is an intervention which involves subjects participating in 9 weekly two-hour therapy groups ('Club meetings') with 3 to 6 other children. The SAS intervention includes a number of components to help children apply the skills that they learn in the session to home. Parents will attend weekly parent support training sessions. 3 and 6 month booster sessions are conducted with both parents and children to help families with maintaining the skills that they have learned and to problem-solve new challenges that arise. Parent and child assessments will be completed at pre and post treatment (Wk 1 and Wk 10) and at 3-month and 6-month follow-up booster visits, for both parent and child participants.
  Interventions: Behavioral: Secret Agent Society (SAS) Program
- Waitlist Group / Treatment As Usual (Other): Participants may be randomly allocated to the wait list control condition, where participants will receive treatment as usual during the 3 month period when the intervention group will participate in the SAS Program. The wait-list group will then be given the opportunity to participate in the SAS intervention at their treating clinic. The wait list control condition includes the treatment participants are already receiving (which may include but is not limited to: individual therapy, group therapy, and/or medication management). Therefore, the wait list control condition consists of treatment which is individually tailored for each participant. Parent and child assessments will be completed at pre and post treatment (Wk 1 and Wk 10) and at 3-month and 6-month follow-up booster visits.
  Interventions: Other: Waitlist Group / Treatment As Usual

INTERVENTIONS:
Behavioral: Secret Agent Society (SAS) Program — The Secret Agent Society (SAS) intervention involves subjects participating in 9 weekly two-hour therapy groups ('Club meetings') with 3 to 6 other children. The SAS intervention includes a number of components to help children apply the skills that they learn in the session to home.
  Arms: Secret Agent Society (SAS) Program
Other: Waitlist Group / Treatment As Usual — The wait list control condition includes the treatment participants are already receiving (which may include but is not limited to: individual therapy, group therapy, and/or medication management). Therefore, the wait list control condition consists of treatment which is individually tailored for each participant. Parent and child assessments will be completed at pre and post treatment (Wk 1 and Wk 10) and at 3-month and 6-month follow-up booster visits. The wait-list group will then be given the opportunity to participate in the SAS intervention at their treating clinic.
  Arms: Waitlist Group / Treatment As Usual

SUMMARY:
Several independent evaluations have supported the effectiveness of the Secret Agent Society (SAS) Program in improving the social-emotional functioning of children with Autism Spectrum Disorders (ASD) in clinic- (Beaumont & Sofronoff, 2008; Tan, Mazzucchelli & Beaumont, submitted), school-(Beaumont, Rotolone & Sofronoff, in press; Einfeld et al., submitted) and remote Skype/telephone-assisted delivery contexts (Sofronoff, Silva & Beaumont, in press).The present study aims to extend on the above literature by conducting a 6-month randomized controlled trial evaluating the effectiveness, utility and acceptability (including cultural acceptability) of the Secret Agent Society (SAS) social-emotional skills training program. Specifically, the study aims to evaluate the effectiveness of the SAS Program for 8-12 year-old children with social difficulties in the context of a range of diagnosed mental health conditions and/or developmental disorders, including anxiety disorders, ADHD, and Autism Spectrum Disorder.

DETAILED DESCRIPTION:
Several independent evaluations have supported the effectiveness of the Secret Agent Society (SAS) Program in improving the social-emotional functioning of children with Autism Spectrum Disorders (ASD) in clinic, school and remote Skype/telephone-assisted delivery contexts. Results from a pilot University clinic evaluation of the program for children with social-emotional difficulties but without ASD has also yielded positive findings, showing comparable treatment effects to those achieved for children with ASD in terms of improved social-emotional functioning. Within the USA, results from a two-year Buffalo School District implementation project and delivery of the program through USC University Center for Excellence in Developmental Disabilities (UCEDD Children's Hospital Los Angeles) have provided further support for the effectiveness and cross-cultural appropriateness of the intervention with children who have a range of mental health challenges. The present study aims to extend on the above literature by conducting a 6-month randomized controlled trial evaluating the effectiveness, utility and acceptability (including cultural acceptability) of the Secret Agent Society (SAS) social-emotional skills training program. Specifically, the study aims to evaluate the effectiveness of the SAS Program for 8-12 year-old children with social difficulties in the context of a range of diagnosed mental health conditions and/or developmental disorders, including anxiety disorders, ADHD, and Autism Spectrum Disorder. Outcome variables will include measures of child social functioning and mental health outcomes related to their primary diagnoses (e.g. anxiety, disruptive behaviour, etc).

ELIGIBILITY:
Inclusion Criteria:

* Children are required to be aged between 8 and 12 years at the time of study entry.
* Children must have a diagnosis of an anxiety disorder, Attention Deficit Hyperactivity disorder and/or Autism Spectrum Disorder and whose parents report that they experience social difficulties/are socially excluded by peers. Participants are not eligible to participate in the study if they do not meet any of the listed diagnoses.
* Children must have an IQ of 85 or above (as formally assessed within the past 2 years, or as assessed at the time of study entry by WIAT III Verbal Subtest).
* Children are required to have significant social difficulties as reported by their parents and/or teacher (although they are not required to score within the clinical range on the Spence Social Skills Questionnaire to be included in the study).
* Children and parents must be fluent in English (preferably their first language).

Exclusion Criteria:

* Failure to meet one or more of the Inclusion Criteria listed above.
* Parents indicate at intake that they are unwilling or unable to attend the parent training sessions and to support their child in completing between-session skills practice tasks ('home missions').
* Children who present with extreme levels of anxiety and anger (as determined from intake interviews and questionnaires), and as such, group therapy would be contraindicated at that time (would cause extreme distress to a child and/or s/he would be a physical safety risk to other child group members).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV-Child Version (ADIS) | 34 weeks. Wk 1, Wk 10, 3-month follow, and 6-month follow-up
  Change in anxiety will be measured at these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bennett, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butterworth TW, Hodge MA, Sofronoff K, Beaumont R, Gray KM, Roberts J, Horstead SK, Clarke KS, Howlin P, Taffe JR, Einfeld SL. Validation of the emotion regulation and social skills questionnaire for young people with autism spectrum disorders. J Autism Dev Disord. 2014 Jul;44(7):1535-45. doi: 10.1007/s10803-013-2014-5. PMID 24337829
- [Result] Beaumont, R., Rotolone, C., & Sofronoff, K. (in press). The Secret Agent Society social skills program for children with a high-functioning autism spectrum disorders: A comparison of two brief versions for schools. Psychology in the Schools. Accepted May 2014.
- [Result] Beaumont R, Sofronoff K. A multi-component social skills intervention for children with Asperger syndrome: the Junior Detective Training Program. J Child Psychol Psychiatry. 2008 Jul;49(7):743-53. doi: 10.1111/j.1469-7610.2008.01920.x. Epub 2008 Jul 1. PMID 18503531
- [Result] Einfeld, S., Sofronoff, K., Gray, K., Roberts, J., Taffe, J., Clark, T., Costley, D., Redoblado Hodge, M.A., Horstead, S., Clarke, K., Beaumont, R., & Howlin, P. (2015). An evaluation of a social skills program for children with autism in specialist schools. Manuscript submitted for publication.
- [Result] Pearson, R., Sofronoff, K., & Beaumont, R. (2015). Preliminary evaluation of the 'Secret Agent Society' social-emotional skills programme with typically developing children. Manuscript in preparation.
- [Result] Sofronoff, K., Silva, J., & Beaumont, R. (2014). Parent delivery of the Secret Agent Society social-emotional skills training program for children with high-functioning autism spectrum disorders. Focus on Autism and Other Developmental Disabilities. Accepted January 2015.
- [Result] Tan, Y.L., Mazzucchelli, T.G., & Beaumont, R. (2015). An evaluation of individually delivered Secret Agent Society social skills program for children with high-functioning autism spectrum disorders: A pilot study. Manuscript submitted for publication.
- [Derived] Temkin AB, Beaumont R, Wkya K, Hariton JR, Flye BL, Sheridan E, Miranda A, Vela J, Zendegui E, Schild J, Gasparro S, Loubriel D, Damianides A, Weisman J, Silvestre A, Yadegar M, Catarozoli C, Bennett SM. Secret Agent Society: A Randomized Controlled Trial of a Transdiagnostic Youth Social Skills Group Treatment. Res Child Adolesc Psychopathol. 2022 Sep;50(9):1107-1119. doi: 10.1007/s10802-022-00919-z. Epub 2022 Apr 20. PMID 35441908